CLINICAL TRIAL: NCT06543563
Title: Esketamine in Microelectrode Recording-guided Subthalamic Deep-Brain Stimulation for Parkinson's Disease（ASPIRE）：A Randomized Controlled, Double-blind Study
Brief Title: Esketamine in Microelectrode Recording-guided Subthalamic Deep-Brain Stimulation for Parkinson's Disease
Acronym: ASPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Director of Anesthesiology Department, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dn20231202
Record Dates: First submitted 2024-07-22; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: PD - Parkinson's Disease; Deep Brain Stimulation; Esketamine
MeSH Terms: conditions — Parkinson Disease | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX (Placebo Comparator): A loading dose of DEX 0.3 µg/kg was infused intravenously at a constant speed within 10 min after the patients entered the operating room, and the DEX maintenance dose was infused at 0.3µg/kg/h until the end of the first stage (deep-brain stimulation implantation) of the operation. After the craniotomy, normal saline is infused at a rate of 3 ml/kg/h until the completion of electrode implantation, prior to microelectrode recording (MER) and electrode insertion. Blood pressure and heart rate of the patient are closely monitored after drug administration to maintain circulatory stability.
  Interventions: Drug: normal Saline
- DEX-KET (Experimental): A loading dose of DEX 0.3 µg/kg was infused intravenously at a constant speed within 10 min after the patients entered the operating room, and the DEX maintenance dose was infused at 0.3µg/kg/h until the end of the first stage (deep-brain stimulation implantation) of the operation. After the craniotomy, esketamine (0.1mg/ml) is infused at a rate of 3ml/kg/h until the completion of electrode implantation, prior to microelectrode recording (MER) and electrode insertion. Blood pressure and heart rate of the patient are closely monitored after drug administration to maintain circulatory stability.
  Interventions: Drug: esketamine

INTERVENTIONS:
Drug: esketamine — After the craniotomy, a continuous infusion of ketamine at a rate of 0.3 mg/kg/h (0.3 ml/kg/h) is administered until the completion of electrode implantation, prior to microelectrode recording (MER) and electrode insertion. After the administration of the drug, close monitoring of the patient's blood pressure and heart rate is conducted to maintain circulatory stability.
  Arms: DEX-KET
Drug: normal Saline — After the craniotomy, a continuous infusion of normal saline at a rate of 0.3 ml/kg/h is administered until the completion of electrode implantation, prior to microelectrode recording (MER) and electrode insertion. After the administration of the drug, close monitoring of the patient's blood pressure and heart rate is conducted to maintain circulatory stability.
  Arms: DEX

SUMMARY:
Under regional anesthesia, subthalamic nucleus deep brain stimulation (STN-DBS) has proven to be an effective therapeutic approach for improving motor symptoms in Parkinson's disease. However, a significant portion of Parkinson's disease (PD) patients is unable to cooperate with the surgery, necessitating the use of awake sedation. Nevertheless, the administration of anesthetic drugs often impacts the electrical signals recorded by microelectrodes to varying degrees. This study is designed as a prospective, randomized, placebo-controlled, double-blind, two-arm investigation. PD patients scheduled for bilateral STN-DBS surgery will be randomly assigned to either the Dexmedetomidine group or the Dexmedetomidine combined with Esketamine group. The differences in neural activity between the two groups will be assessed using the normalized root mean square (NRMS) method. The primary outcome measure is NRMS, while secondary outcome measures include differences in beta oscillation power spectrum analysis, postoperative delirium incidence, postoperative changes in sleep disturbances, postoperative depression, anxiety status, and occurrence of adverse events.

DETAILED DESCRIPTION:
Regional anesthesia for subthalamic nucleus deep brain stimulation (STN-DBS) is an effective treatment method for improving motor symptoms in Parkinson's disease. However, the majority of Parkinson's disease (PD) patients require awake sedation during the procedure. Nevertheless, the administration of anesthetic drugs often impacts the microelectrode recording (MER) signals to varying degrees. Current research suggests that Esketamine can provide sedation and analgesia while preserving the active brain electrical signals of patients. Additionally, it has been shown to improve sleep disturbances and alleviate depression and anxiety in patients.This study aims to compare the impact of Dexmedetomidine alone and Dexmedetomidine combined with Esketamine on MER during awake sedation in PD patients undergoing STN-DBS surgery, to clarify the influence of Esketamine on the intraoperative electrical signals of PD patients under awake sedation during DBS surgery. The experiment is designed as a prospective, randomized, placebo-controlled, non-inferiority study with a double-blind, two-arm design. PD patients scheduled for bilateral STN-DBS surgery will be randomly assigned to either the Dexmedetomidine group or the Dexmedetomidine combined with Esketamine group. The differences in neural activity between the two groups will be assessed using the normalized root mean square (NRMS) method. The primary outcome measure is NRMS, while secondary outcome measures include differences in beta oscillation power spectrum analysis, postoperative delirium incidence, postoperative changes in sleep disturbances, postoperative depression, anxiety status, and occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1.50-80 years old, ASA grade II-III; 2.Bilateral STN-DBS of patients with Parkinson's disease; 3.Signed informed consent.

Exclusion Criteria:

1. Obstructive sleep apnea;
2. BMI > 30kg/m2;
3. Estimated difficult airway;
4. Severe preoperative anxiety;
5. Serious dysfunction of important organs (i.e. heart failure, renal or liver dysfunction)
6. A history of allergy to the anaesthetics.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-08-09 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
NRMS | 1 day (during MER recording)
  The investigators will use the root mean square (RMS) value of the MER sampled signal as the main parameter for evaluating electrode position. RMS values change with the electrode properties and other external drives related to the operating room; therefore, it is crucial to normalize the RMS to comparable values. Thus, each session's RMS in a trajectory is divided by the mean RMS of the first five stable sessions in the same trajectory. This normalized RMS (NRMS) is found to be a good measure as it reflects the relative change in the total power of the signal, which elevates dramatically entering the STN.

SECONDARY OUTCOMES:
Beta band (13-30 Hz) oscillations calculated by spectrum analysis | 1 day (during MER recording)
  Power spectrum will be calculated using a discrete Fourier transform of the sampling windows to allow evaluation of change in oscillatory activity along time. Synchronized beta band (13-30 Hz) oscillations are often observed in the dorsolateral region of the STN of PD patients and are thought to play a role in the disease pathophysiology. The power of beta band will be calculated by averaging the power across the corresponding frequency band.
Early postoperative Quality of sleep | the first and the second and the third day after surgery
  The early postoperative sleep quality will be monitored using a portable sleep monitor, with indicators including the duration of total sleep, the proportion of light sleep, deep sleep, and rapid eye movement (REM) sleep.
Long-term Quality of sleep | before surgery and the 30days after surgery
  Long-term quality of sleep will be evaluated with Pittsburgh Sleep Quality Index (PSQI) ,a score of 0 to 21, the higher score means a worse quality of sleep.
Anxiety | before surgery and the 30days after surgery
  Anxiety will be evaluated using Hamilton Anxiety Rating Scale (HAMA)，a score of 0 to 56，the higher score means a worse anxiety
Depression | before surgery and the 30days after surgery
  Depression will be evaluated using Hamilton Depression Rating Scale (HAMD)，a score of 0 to 76,the higher score means a worse depression
Delirium Assessment: 3-Minute Diagnostic Interview for CAM (3D-CAM) | Postoperative 3 days and the 30th day
  Postoperative delirium is assessed by the 3-minute diagnostic interview for CAM(3D-CAM),the score is 0 or 1, where 0 represents non-delirium and 1 represents delirium.
The incidence of anaesthesia-related adverse events | Up to 3 days after randomization]
  Nausea, vomiting, excessive Secretions and intraoperative awareness
Surgical experience satisfaction 24 hours after the operation and DBS satisfaction 1 months after the operationevaluated by the seven-point Likert scale | 24 hours after operation for surgical experience satisfaction and 1 months after STN-DBS for DBS satisfaction
  The seven-point Likert scale will be used in the present trial. It is a questionnaire answered by the patient 24 hoursafter the operation. The scale reported the experience of the patient from very dissatisfied to very satisfied, as graded from 1-7.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, MD,PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR